CLINICAL TRIAL: NCT03238339
Title: The Clinical Application and Popularization of Portable Home Noninvasive Ventilator
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mingdong Hu (Other)
Responsible Party: Sponsor-Investigator, Mingdong Hu, associate chief physician, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: cstc2016shmszx130034
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Hypercapnic Respiratory Failure
Keywords: Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Oxygen Inhalation Therapy; Noninvasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Portable Home Noninvasive Ventilator treatment group: The patients maintain a stable COPD regimen, and on the basis of conventional home oxygen therapy, a portable, wearable, non-invasive ventilator will be used.
- Routine home oxygen therapy group: The patient maintained a stable COPD regimen and conventional home oxygen therapy.

SUMMARY:
The subjects of this study are the chronic obstructive pulmonary disease (COPD) patients with chronic II respiratory failure. The participants will be divided into two groups: The Portable Home Noninvasive Ventilator treatment group and the routine home oxygen inhalation treatment group. All subjects will be given a stable COPD regimen and conventional oxygen therapy ,but the portable home noninvasive ventilator treatment group will need to wear a portable non-invasive ventilator. Objective evaluation indexes were established during the routine treatment, and two groups of subjects will be followed up for one year. Finally, the clinical data of all subjects will be analyzed，and then the practicability of portable wearable household noninvasive ventilator will be verified.The researchers will also build a remote breathing data-monitoring platform based on mobile internet,and a community home demonstration application point.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old < age < 80 years old
* COPD diagnosis was made according to GOLD guidelines
* The subjects with chronic type II respiratory failure
* The subjects with structural lung disease
* The subjects signed informed consent.

Exclusion Criteria:

* The subjects suffering from COPD acute exacerbation
* The subjects currently participating in other related products
* The subjects with organ dysfunction because of liver,kidney, hematopoietic system and serious metabolic disease endocrine system
* The subjects with poor compliance
* The subjects refused to sign the informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects were selected from the Department of respiration, Xinqiao Hospital of Chongqing city.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of the chronic obstructive pulmonary disease(COPD) acute exacerbation. | one year
  Record the frequency of COPD acute exacerbation within one year

SECONDARY OUTCOMES:
The first onset time of the chronic obstructive pulmonary disease(COPD) acute exacerbation | one year
  Record the first onset time of COPD acute exacerbation
The number of hospitalizations due to the chronic obstructive pulmonary disease(COPD) acute exacerbation | one year
  Record the number of hospitalizations due to the COPD acute exacerbation

OTHER OUTCOMES:
Six Minute Walk Distance | month0,month4,month8,month12
pulmonary arterial pressure | month0,month4,month8,month12
arterial blood gas | month0,month4,month8,month12
routine analysis of blood | month0,month4,month8,month12
The change of cytokines expression | month0,month4,month8,month12
  The cytokines including IL8、IL13、TNF-a、INF-r、IFN-γ、LTB4.

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department, Xinqiao Hospital, Third Military Medical University, Chongqing, China